CLINICAL TRIAL: NCT02144896
Title: Ankle Dorsiflexion Splinting Enhances Endothelial Function of Aged Leg Muscles
Brief Title: Effect of Ankle Splinting on Vascular Function in Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 122-2013-N; 1R21AG044858-01A1 (NIH)
Record Dates: First submitted 2014-05-15; First posted 2014-05-22 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Aging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ankle splinting (Experimental): Older adults will have one leg randomly assigned to ankle splinting for 4 weeks. The non-splinted leg will serve as the control.
  Interventions: Other: Ankle splinting
- No Ankle Splinting (No Intervention): The non splinted leg will serve as the control

INTERVENTIONS:
Other: Ankle splinting — Ankle dorsiflexion splinting will be performed 30 minutes per day, 5 days per week for 4 weeks.
  Arms: Ankle splinting

SUMMARY:
Endothelial function of the skeletal muscle vasculature declines with advancing age. Although aerobic exercise training is commonly prescribed to combat loss of endothelial function in the elderly, the rate of compliance to training programs is low. Contrary to aerobic exercise training, stretching exercise is widely performed in elderly patients to increase muscle flexibility and to prevent muscle atrophy induced by immobilization. However, it remains unknown as to whether regular stretching of the calf muscles using ankle dorsiflexion splinting improves muscle blood flow. The purpose of the proposed work is to test the hypothesis that performance of ankle dorsiflexion splinting improves endothelial function and lower leg muscle blood flow in older adults. Ankle dorsiflexion splinting will be performed on the randomized leg for 30 minutes, 5 times per week for 4 weeks. Leg vascular measures will be performed on the splinted and non-splinted legs prior to and at the end of the 4-week intervention.

DETAILED DESCRIPTION:
Older adults will be recruited in this study. Vascular function will be assessed before and after the 4-week ankle splinting intervention. To examine the acute effects of splinting, vascular measures will also be obtained before and immediately following 30 min of ankle splinting. All procedures will be performed at the Integrative Cardiovascular Physiology Laboratory at the University of Florida.

Participants will have one leg randomly assigned to using a splint to stretch the calf muscles 30 min per day, 5 days per week for 4 weeks, while the contralateral non-splinted leg will serve as an internal control.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 60 to 79 years.
* Women will all be postmenopausal and must not take hormone replacement therapy.
* Sedentary, defined as no regular exercise training.

Exclusion Criteria:

* No evidence of heart disease evidenced by abnormal resting ECG, angina or ECG evidence of acute myocardial ischemia during the exercise test, no history of any relevant acute cardiac event (myocardial infarction, episode of heart failure)
* No history of deep vein thrombosis.
* No history of Type I or II diabetes mellitus.
* No history for renal or liver disease.
* No history of seizures, or other relevant on-going or recurrent illness.

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-04-10 (Actual); Study Completion 2015-04-10 (Actual)

PRIMARY OUTCOMES:
Change in vascular endothelial function of leg conduit artery | At baseline and after 4 weeks of ankle splinting
  Endothelium-dependent and endothelium-independent dilation of popliteal artery using ultrasonography.

SECONDARY OUTCOMES:
Change in vascular endothelial function of calf resistance vessels | At baseline and after 4 weeks of ankle splinting
  Vascular endothelial function of calf resistance vessels using venous occlusion plethysmography.
Change in calf blood flow in response to acute ankle splinting | Before and after 30 min of ankle splinting
  Calf blood flow using ultrasonography and venous occlusion plethysmography before and after acute splinting.

CONTACTS AND LOCATIONS:
Overall Officials: Demetra D Christou, Ph.D, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No